CLINICAL TRIAL: NCT01407705
Title: High-Resolution Diffusion Tensor Imaging (DTI) of the Cervical Spinal Cord in the Setting of Spinal Cord Injury (SCI)
Status: Completed | Type: Observational
Sponsor: University of Utah (Other)
Responsible Party: Principal Investigator, Brandon Lawrence, M.D., University of Utah
Other Study IDs: 22962
Record Dates: First submitted 2011-07-29; First posted 2011-08-02 (Estimated); Last update posted 2014-05-21 (Estimated); Status verified 2014-05

CONDITIONS: Spinal Cord Injury; Cervical Spondylosis With Myelopathy; Degenerative Disorder
Keywords: spinal cord injury with traumatic event
MeSH Terms: conditions — Spinal Cord Injuries

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (2):
- Control Group: * No diagnosis of cervical degenerative or traumatic disease
  * 30 to 80 years of age
  * Ability of volunteers to tolerate 1 hr examination
- Disease (Non-healthy) Group: Cervical Spinal Cord:
  * Clinical and Radiographic evidence of cervical spondylotic myelopathy
  * 18 to 80 years of age
  * Safe and stable clinical scenario to undergo imaging
  * Awake, alert patient able to cooperate with physical examination
  * Give written informed consent prior to any testing under this protocol
  Degenerative Disease Group:
  * Have signs or symptoms consistent with spinal cord injury.
  * Be diagnosed with cervical spondylosis (degenerative disease).
  Traumatic Group:
  • A spinal cord injury associated with a traumatic event.

SUMMARY:
The investigators propose a prospective study, designed to analyze the efficacy of High-Resolution Diffusion Tensor Imaging for accurately sensing white matter tracts in subjects with spinal cord injury. Study subjects will not be randomized, as treatment will follow the doctor's "standard of care." Patients will be selected and offered enrollment based upon the clinical diagnosis of spinal cord injury, either due to degenerative disease or trauma. Enrollment will be based on the chronology of patient presentation.

DETAILED DESCRIPTION:
Spinal cord injury (SCI) can result from trauma as well as degenerative conditions, such as cervical spondylotic myelopathy (CSM). Both have a profound impact on the physical and mental health of the affected individual. The symptoms of CSM can include weakness in the arms or legs, difficulty with walking and balance, loss of dexterity in the hands, and bowel or bladder dysfunction. Traumatic spinal cord injury often includes damage to white matter tracts resulting in irreversible functional deficits such as paraplegia or quadriplegia.

Although current diagnostic imaging can reveal highly specific parameters of spinal canal anatomy, the functional anatomy of the spinal cord remains unknown. Patients with similar diagnostic findings can vary clinically with many patients having minimal to no symptoms while others may be severely incapacitated. Conventional MRI methods, such as T1/T2 weighted MRI, may easily identify the region of the damage and may depict permanent changes in the spinal cord tissue. However, conventional MRI methods are limited in their ability to correlate imaging findings with short and long term functional outcomes from spinal cord injury. DTI has the potential to improve upon conventional MRI imaging by providing information about tissue microstructure and may be particularly well suited for assessing the integrity of fiber tracts in SCI.

Diffusion tensor magnetic resonance imaging (DTI) is a new technique that is highly sensitive in detecting the integrity of white matter tracts. Although information obtained from DTI has been utilized for white matter abnormalities in the brain, DTI of the spinal cord in vivo has provided many challenges. The small size of the spinal cord and the close packing of its white matter tracts require a very high image resolution to visualize these individual tracts. The resolution required to image the small cross sectional area of the spinal cord has been difficult to achieve using most widely used DTI sequences. To date, DTI measurements reports have demonstrated a practical application of DTI on the cervical spinal cord with limited spatial resolutions from 8 mm3 to 16 mm3.

To achieve high-resolution DTI of the spinal cord, two novel imaging techniques for high-resolution in-vivo DTI on a clinical 3T MRI system (Trio, Siemens Medical Solution, Erlangen Germany) have been developed: 2D singleshot Interleaved Multiple Inner Volume DWEPI (ss-IMIV-DWEPI) and 3D singleshot DW STimulated EPI (3D ss-DWSTEPI). These optimized DTI pulse sequences have typically achieved approximately 2.0 or 1.253 mm3 spatial resolution within clinically achievable imaging time (~5 min.). The sequences have been designed especially for high-resolution DTI of cervical spinal cord. They have been applied to spinal cord specimens ex vivo as well as to a small group of healthy volunteers and multiple sclerosis patients.

ELIGIBILITY:
Inclusion Criteria:

* For inclusion to the Cervical Spinal Cord (CSM)

  * Clinical and Radiographic evidence of cervical spondylotic myelopathy
  * 18 to 80 years of age
  * Safe and stable clinical scenario to undergo imaging
  * Awake, alert patient able to cooperate with physical examination
  * Give written informed consent prior to any testing under this protocol

For inclusion to the Control Group, subject must have:

* No diagnosis of cervical degenerative or traumatic disease
* 30 to 80 years of age
* Ability of volunteers to tolerate 1 hr examination

For inclusion to the Degenerative Disease Group, subject must:

* Have signs or symptoms consistent with spinal cord injury.
* Be diagnosed with cervical spondylosis (degenerative disease).

For inclusion to the Traumatic Group, subject must have:

• A spinal cord injury associated with a traumatic event.

Exclusion Criteria:

* For exclusion to the Cervical Spinal Cord (CSM):

  * Unsafe or unstable clinical scenario
  * Prior cervical spine surgery
  * History of neurological disease (stroke, multiple sclerosis, peripheral neuropathy, or other neurodegenerative conditions)
  * Inability to comply with physical examination
  * Contraindications to MRI imaging (metal debris, cardiac pacemaker, etc..)
  * Pregnant women

For exclusion to the other groups:

* Inability to comply with physical examination
* Contraindications to MRI imaging (metal debris, cardiac pacemaker, etc..)
* Pregnant women

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Study subjects will not be randomized, as treatment will follow the doctor's "standard of care." Patients will be selected and offered enrollment based upon the clinical diagnosis of spinal cord injury, either due to degenerative disease or trauma. Enrollment will be based on the chronology of patient presentation.
Sampling Method: Non-Probability Sample
Enrollment: 31 (Actual)
Dates: Start 2007-05; Primary Completion 2014-05 (Actual); Study Completion 2014-05 (Actual)

PRIMARY OUTCOMES:
high-resolution DTI of cervical spinal cord | 2 years
  To determine the efficacy of high-resolution diffusion weighted pulse sequence with spatial resolution of 2.0 mm3 to confirm directionality and intactness of cervical spinal cord tracts in vivo in the setting of spinal cord injury and disease-free subjects.

CONTACTS AND LOCATIONS:
Overall Officials: Brandon Lawrence, MD, Principal Investigator — University of Utah Orthopedics
Locations (1):
- University of Utah Orthopedics, Salt Lake City, Utah, United States